CLINICAL TRIAL: NCT06710418
Title: Red Blood Cell Transfusion Threshold-Specific Bleeding, Quality of Life and Functional Outcomes in Acute Leukemia Patients With Thrombocytopenia: a Randomized Feasibility Study
Brief Title: Evaluating the Effects of Hemoglobin Threshold-specific Packed Red Blood Cell Transfusions on Quality of Life and Functional Outcomes in Patients With High-grade Myeloid Neoplasms, Acute Myeloid Leukemia, or B Acute Lymphoblastic Lymphoma/Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1124891; NCI-2024-09018 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20807 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-11-14; First posted 2024-11-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Myeloid Leukemia; B Acute Lymphoblastic Leukemia; B Lymphoblastic Lymphoma; Myeloid Neoplasm
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Burkitt Lymphoma; Precursor B-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Specimen Handling; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (restrictive threshold) (Experimental): Patients undergo PRBC transfusion if at any point their hemoglobin level is 7 gm/dL or less, starting the day after SOC chemotherapy/stem cell infusion is complete and continuing for up to 42 days. Patients also undergo collection of blood samples on study.
  Interventions: Other: Activity Tracking; Procedure: Biospecimen Collection; Procedure: Cognitive Assessment; Other: Electronic Health Record Review; Other: Packed Red Blood Cell Transfusion; Other: Quality-of-Life Assessment
- Arm II (liberal threshold) (Experimental): Patients undergo PRBC transfusion if at any point their hemoglobin level is 9 gm/dL or less, starting the day after SOC chemotherapy/stem cell infusion is complete and continuing for up to 42 days. Patients also undergo collection of blood samples on study.
  Interventions: Other: Activity Tracking; Procedure: Biospecimen Collection; Procedure: Cognitive Assessment; Other: Electronic Health Record Review; Other: Packed Red Blood Cell Transfusion; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Activity Tracking — Ancillary studies
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Cognitive Assessment — Ancillary studies
Other: Electronic Health Record Review — Ancillary studies
Other: Packed Red Blood Cell Transfusion — Undergo PRBC transfusion
  Other Names: PRBC Transfusion
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This clinical trial evaluates the effects of hemoglobin threshold-specific packed red blood cell (PRBC) transfusions on quality of life and functional outcomes in patients who have undergone chemotherapy or an allogeneic hematopoietic stem cell transplant for a high-grade myeloid neoplasm, acute myeloid leukemia, or B acute lymphoblastic lymphoma/leukemia. Some types of chemotherapy and stem cell transplants can induce low platelet counts and/or anemia that requires PRBC transfusions. Given critical shortages in blood supply, and risks associated with transfusion of PRBC, there has been much investigation into the "minimum" hemoglobin level that effectively balances safety and toxicity in patients. This clinical trial evaluates the effects of giving PRBC transfusions based on a more restrictive hemoglobin threshold (> 7 gm/dL) compared to a more liberal hemoglobin threshold (> 9 gm/dL) on quality of life and functional outcomes. A more restrictive threshold may be just as effective at maintaining patient quality of life and function while decreasing side effects from blood transfusions and helping to conserve blood supply resources.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo PRBC transfusion if at any point their hemoglobin level is 7 gm/dL or less, starting the day after standard of care (SOC) chemotherapy/stem cell infusion is complete and continuing for up to 42 days. Patients also undergo collection of blood samples on study.

ARM II: Patients undergo PRBC transfusion if at any point their hemoglobin level is 9 gm/dL or less, starting the day after SOC chemotherapy/stem cell infusion is complete and continuing for up to 42 days. Patients also undergo collection of blood samples on study.

After completion of study intervention, patients are followed up for 7 days and then periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of "high-grade" myeloid neoplasm (≥ 10% blasts in blood or bone marrow) or acute myeloid leukemia (AML) (other than acute promyelocytic leukemia [APL]) or B-cell acute lymphoblastic lymphoma/leukemia (ALL) according to the 2022 WHO classification. Outside diagnostic material is acceptable to establish diagnosis
* Plan to undergo intensive chemotherapy induction or post-remission therapy for their diagnosis (defined as "7+3," hyper-cyclophosphamide, vincristine, doxorubicin, and dexamethasone [CVAD], or regimen with cytarabine backbone ≥ 1,000mg/m^2), or allogeneic HSCT, expected to induce anemia requiring PRBC transfusion AND platelet counts of ≤ 30,000/uL for ≥ 5 days following the therapy (as determined by principal investigator)
* Plan to get all post-chemotherapy/post-HSCT care at the University of Washington (UW)/Fred Hutchinson Cancer Center (FHCC)
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients requiring a prophylactic platelet transfusion at thresholds > 10,000/uL
* Patients requiring systemic anticoagulation, anti-platelet agent, or antifibrinolytic therapy that will not be held once platelets reach a level of < 50,000/uL
* Patients with grade ≥ 2 bleeding (as determined by the WHO Bleeding Criteria) at the time of randomization
* Arterial or venous thrombotic event, including myocardial infarction within 6 months prior to initiation of the chemotherapy/HSCT
* Patients requiring renal replacement therapy at the time of randomization
* Patients who decline transfusion for personal or religious beliefs
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible patients that consent (feasibility) | Up to 30 months
  Randomizing patients to two different transfusion thresholds will be considered feasible if greater than 50% of eligible patients consent.
Percentage of patients randomized to the restrictive 7 gm/dL threshold that tolerate this transfusion trigger (feasibility) | Up to 7 days after completion of study intervention
  Randomizing patients to two different transfusion thresholds will be considered feasible if greater than 75% of the patients randomized to the restrictive 7 gm/dL threshold tolerate this transfusion trigger. A patient will be defined as tolerant if the patient receives transfusions at a hemoglobin threshold higher than > 7gm/dL less than 3 times due to signs/symptoms of acute anemia.
Indication for early termination based on interim analyses of safety (feasibility) | Up to 30 months
  Randomizing patients to two different transfusion thresholds will be considered feasible if there is no indication for early termination based on the interim safety analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Halpern, MD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No